CLINICAL TRIAL: NCT03046459
Title: A First-in-human Study to Characterize the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of BNZ132-1-40
Brief Title: A First-in-Human Study of BNZ132-1-40
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioniz Therapeutics (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BNZ-CT-101
Record Dates: First submitted 2017-01-25; First posted 2017-02-08 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: cytokines; interleukin-2; Safety Issues

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BNZ132-1-40 (Experimental): a range of IV doses
  Interventions: Biological: BNZ132-1-40

INTERVENTIONS:
Biological: BNZ132-1-40 — pegylated peptide inhibiting IL-2, IL-9 and IL-15

SUMMARY:
This is an open-label, single ascending dose study to characterize the safety and PK/PD profile of IV BNZ132-1-40, a novel peptide inhibitor of multiple cytokines in the IL-2 family.

DETAILED DESCRIPTION:
This is a open-label study of single doses of intravenous BNZ132-1-40 administered to healthy adult subjects. Subjects are followed for 30 days after treatment for collection of safety, PK and PD data. Cohorts of up to 6 subjects will be enrolled for each dose level.

ELIGIBILITY:
Inclusion Criteria:

* males and non-pregnant, non-lactating females
* no ongoing clinically significant medical condition
* willing and able to provide informed consent
* no use of Rx or OTC medications, other than oral contraceptives

Exclusion Criteria:

* Recent systemic infections
* Clinically-significant abnormal clinical labs, ECG or physical examination
* Immunization 30 days prior to study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with related, treatment-emergent adverse events | 30 days

SECONDARY OUTCOMES:
PK: Exposure as determined by maximum plasma concentration (Cmax) | 1 Day
PK: Exposure as determined by area under the concentration-time curve (AUC) | 30 days
PD: Effects of BNZ132-1-40 on the expression of T cells as determined by FACS analysis | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Frohna, MD, PhD, Study Director — Bioniz Therapeutics, Inc.
Locations (1):
- Celerion, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nata T, Basheer A, Cocchi F, van Besien R, Massoud R, Jacobson S, Azimi N, Tagaya Y. Targeting the binding interface on a shared receptor subunit of a cytokine family enables the inhibition of multiple member cytokines with selectable target spectrum. J Biol Chem. 2015 Sep 11;290(37):22338-51. doi: 10.1074/jbc.M115.661074. Epub 2015 Jul 16. PMID 26183780